CLINICAL TRIAL: NCT05901415
Title: Combined Anterior Lumbar Plexus and Lateral Sacral Plexus Block in a Semi-supine Position for Hip Fracture Surgery in Elderly Patients: A Randomized Controlled Trial
Brief Title: Modified LPB and SPB vs Classical LPB and SPB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K3105
Record Dates: First submitted 2023-04-17; First posted 2023-06-13 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: A modified semi-supine position of combined anterior lumbar and lateral sacral plexus block
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Modified Semi-supine Position of Combined Anterior Lumbar and Lateral Sacral Plexus Block (Experimental): Patients were placed in a supine position with a small pad put under the upper body at the surgical side, then they received a combined anterior lumbar and lateral sacral plexus block.
  Interventions: Procedure: Combined anterior lumbar plexus and lateral sacral plexus block in a semi-supine position
- A classical Position of Combined Anterior Lumbar and Lateral Sacral Plexus Block (Sham Comparator): Patients received a combined anterior lumbar and lateral sacral plexus block in a lateral position.
  Interventions: Procedure: Combined anterior lumbar plexus and lateral sacral plexus block in a classical position.

INTERVENTIONS:
Procedure: Combined anterior lumbar plexus and lateral sacral plexus block in a semi-supine position — We proposed a modified approach of combined anterior LPB and lateral SPB with the patients posed in a semi-supine position aiming to reduce the pain and discomfort induced by position changing effectively.
  Arms: A Modified Semi-supine Position of Combined Anterior Lumbar and Lateral Sacral Plexus Block
Procedure: Combined anterior lumbar plexus and lateral sacral plexus block in a classical position. — Patients posed in a classical position and received combined anterior LPB and lateral SPB.
  Arms: A classical Position of Combined Anterior Lumbar and Lateral Sacral Plexus Block

SUMMARY:
The timing of surgery for hip fractures is crucial for elderly patients. The mortality rate for elderly patients after hip fracture is high, and anesthetic decisions significantly affect the patient's outcome. Regional anesthesia has been shown to have better outcomes than general anesthesia. We proposed a newly developed modified position for the ultrasound-guided combined anterior lumbar and lateral sacral plexus block technique that offers benefits, including minimizing interference with circulation and anesthesia, avoiding position change and pain, and providing effective postoperative analgesia.

DETAILED DESCRIPTION:
The increasing proportion of elderly patients requiring surgery, particularly for hip fractures, is common among the elderly. The timing of surgery for hip fractures is crucial and most require surgical treatment. The mortality rate for elderly patients after hip fracture is high, and anesthetic decisions significantly affect the patient's outcome. Elderly patients have decreased physiological function and are more susceptible to postoperative complications, such as delirium, constipation, pressure sores, and catheter-related infections. Regional anesthesia has been shown to have better outcomes than general anesthesia. We proposed a newly developed modified position for the ultrasound-guided combined anterior lumbar and lateral sacral plexus block that offers benefits, including minimizing interference with circulation and anesthesia, avoiding position change and pain, and providing effective postoperative analgesia. The study validates the feasibility and effectiveness of this technique for elderly hip fracture surgery and compares it with a traditional lumbar-sacral plexus nerve block, providing a fresh perspective on anesthesia for this type of surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients over 70 years of age. ASA classification grades II-IV. Patients with hip fractures requiring surgery (intramedullary nailing of intertrochanteric fractures).

Exclusion Criteria:

Peripheral neuropathy or other neurological disorders affecting the nerves involved in the block; Serve coagulopathy or platelet dysfunction; Inability to perform puncture due to infection, wound, or other reasons at the puncture site; Allergy to local anesthetics or any other medications used in the block; Inability to cooperate or communicate with the healthcare provider during the procedure; Patients or their families who cannot understand the conditions and objectives of the study.

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale Score | up to 3 months
  Compared VAS score of two approaches in patients undergoing anesthesia（VAS from the minimum 0 to the maximum 10 scores）

CONTACTS AND LOCATIONS:
Overall Officials: Xulei Cui, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Heyu Ji, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ji H, Cui X. A modified approach of combined anterior lumbar plexus block with lateral sacral plexus block in a semi lateral supine position for lower limb fracture patients: a case series. BMC Anesthesiol. 2025 Feb 14;25(1):74. doi: 10.1186/s12871-025-02943-0. PMID 39953416